CLINICAL TRIAL: NCT01766947
Title: A Prospective, Open Label Study to Assess the 24-hour Intraocular Pressure Fluctuation Profile Recorded With SENSIMED Triggerfish® in Patients With Primary Open Angle Glaucoma Before and After Deep Sclerectomy
Brief Title: IOP Fluctuations in Primary Open Angle Glaucoma Patients Before and After Deep Sclerectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TF-1206
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Glaucoma; Deep sclerectomy
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triggerfish (Experimental): Device : Sensimed Triggerfish
  Interventions: Device: Sensimed Triggerfish

INTERVENTIONS:
Device: Sensimed Triggerfish — Portable investigational device using a contact lens sensor that monitors the IOP fluctuation continuously over 24-hours

SUMMARY:
Primary open angle glaucoma (POAG) is associated with inadequate drainage of the aqueous humor via the trabecular meshwork through the Schlemm's canal towards the systemic circulation. This may lead to an increase in IOP and may damage the optic nerve. The purpose of glaucoma management is to lower IOP in order to prevent progression of the optic neuropathy and subsequent visual loss. Firstline treatment usually includes IOP-lowering drug therapy. However, if IOP remains uncontrolled and/or the optic nerve damage progresses despite controlled IOP, surgery may be indicated. Deep sclerectomy (DS) is a non-penetrating surgical procedure for the treatment of open angle glaucoma that allows the enhancement of the aqueous outflow by removing part of the inner wall of Schlemm's canal and trabecular meshwork. DS was shown to achieve a good control on IOP over the long term.

The purpose of this study is to assess the 24-hour IOP fluctuation profile recorded with Triggerfish in patients with POAG before and after DS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of POAG
* Documented glaucomatous VF damage with mean defect (MD) > 3 dB
* Progressing glaucomatous damage justifying a DS
* Aged ≥18 years, of either sex
* Not more than 4 diopters spherical equivalent on the study eye
* Not more than 2 diopters cylinder equivalent on the study eye
* Have given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* Corneal or conjunctival abnormality precluding contact lens adaptation
* Severe dry eye syndrome
* Patients with allergy to corneal anesthetic
* Patients with contraindications for silicone contact lens wear
* Patients not able to understand the character and individual consequences of the investigation
* Participation in other clinical research within the last 4 weeks
* Any other contra-indication listed in the Triggerfish user manual

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Effect of DS on IOP fluctuation profile as recorded by Triggerfish in patients with POAG. | 3 months
  The IOP fluctuation profile will be recorded by Triggerfish in patient with POAG
  * Before DS
  * 3 months after DS

SECONDARY OUTCOMES:
effect of DS on the diurnal and nocturnal IOP fluctuation pattern | 3 months
  Diurnal and nocturnal IOP fluctuation pattern The wake/sleep and sleep/wake Triggerfish slopes Timing of Triggerfish acrophase
Changes in visual field up to 6 months after DS | 3 months
  Change in the visual field
Safety and Tolerability | 3 months
  Adverse events and serious adverse events will be collected throughout the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Baudouin, MD, Principal Investigator — Centre hosptilatier National d'Opthalmologie des Quinze-Vingts
Locations (1):
- Centre Hospitalier National d'Opthalmology des Quinze-Vingts, Paris, France